CLINICAL TRIAL: NCT06737406
Title: Efficacy and Safety of 5-Fluorouracil (5FU) in Combination With Calcipotriol in Children (Aged 4 to 18 Years) With Palmoplantar Wart: Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Topical 5-Fluorouracil (5FU) Plus Calcipotriol in Children With Palmoplantar Wart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Malekan, Medical Doctor, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.MAZUMS.REC.1403.120
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Common Warts
Keywords: Wart; 5-Fluorouracil; Calcipotriol; Children
MeSH Terms: conditions — Warts

STUDY DESIGN:
Intervention Model Description: This study will be a single-center, parallel, randomized, double-blind, placebo-controlled trial. Patients who meet eligibility criteria will be randomized (1:1:1) to one of 3 groups. Group A will receive 5% fluorouracil cream and 0.005% calcipotriol ointment. Group B will receive 5% fluorouracil cream and a placebo ointment in identical tubes in terms of color and scent and with identical usage instructions to calcipotriol. Group C will receive 0.005% calcipotriol ointment and a placebo cream in identical tubes with identical instructions to fluorouracil. All patients applied a thin layer of ointment and cream to the affected area (palmoplantar) twice daily for 3 consecutive weeks (21 days).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): 5% fluorouracil cream + 0.005% calcipotriol ointment
  Interventions: Drug: Topical 5% fluorouracil cream; Drug: Topical 0.005% calcipotriol ointment
- B (Experimental): 5% fluorouracil cream + Placebo
  Interventions: Drug: Topical 5% fluorouracil cream; Drug: Placebo
- C (Experimental): 0.005% calcipotriol ointment + Placebo
  Interventions: Drug: Topical 0.005% calcipotriol ointment; Drug: Placebo

INTERVENTIONS:
Drug: Topical 5% fluorouracil cream — Topical 5% fluorouracil cream twice daily for 21 days on the affected area (palmoplantar)
  Arms: A; B
Drug: Topical 0.005% calcipotriol ointment — Topical 0.005% calcipotriol ointment twice daily for 21 days on the affected area (palmoplatar)
  Arms: A; C
Drug: Placebo — A placebo ointment in identical tubes in terms of color and scent and with identical usage instructions to calcipotriol.
  Arms: B
Drug: Placebo — A placebo cream in identical tubes in terms of color and scent and with identical usage instructions to fluorouracil.
  Arms: C

SUMMARY:
Warts caused by the human papillomavirus (HPV) are one of the most common skin conditions among children. The prevalence of warts in school-aged children ranges from 10 to 20 percent. Warts are more common among immunocompromised patients [1, 2]. Some studies also show that the prevalence of viral warts in the pediatric population increases with age, peaking in adolescence. HPV is a DNA virus that replicates only in fully differentiated epithelial cells. More than 80 types of HPV have been identified. Types 27, 57, 2, and 1 are the most common types of HPV in skin warts in the general population. Warts usually affect patients of different age groups and various parts of the body, causing physical and psychological complications for patients (such as pain, discomfort, and embarrassment), which in turn lead to functional impairment. Warts often affect pressure points on the soles of the feet. Although most warts are asymptomatic, plantar warts are often associated with pain while walking, causing physical and psychological stress [3].

Various treatments such as keratolytic agents, cryotherapy, laser, antimitotic treatments, contact sensitizers, and intralesional injection of antigen have been used. There is no evidence that one treatment is superior to others, and in many cases, treatment of viral warts requires a combination of treatments. Treatment selection for patients should be based on variables such as wart size, number of lesions, anatomical location, patient preference, cost, convenience, side effects, and operator experience. It is important to emphasize that good communication between the patient, parents, and dermatologist is essential for successful treatment in children [2, 4].

Despite having various treatment approaches, treating plantar warts is challenging. No single treatment is effective in most patients, treatments are often painful, and they are associated with a high recurrence rate. Although nearly 75 percent of warts can resolve spontaneously within two years, patients often seek treatment for cosmetic reasons and pain. Many studies have examined the use of vitamin D compounds (calcipotriol) and 5-fluorouracil in wart patients separately or in combination with other drugs, but only one recent case report that tested the combination of these two showed very positive efficacy results [5, 6].

To date, no clinical trial has evaluated the combination of calcipotriol and 5-fluorouracil. Additionally, given that common current treatments such as cryotherapy are painful for children, achieving an effective, pain-free intervention is necessary. This study aims to evaluate the efficacy and side effects of the combination of 5-fluorouracil and calcipotriol in children (ages 4 to 18) with palmar and plantar warts in a randomized, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria include the clinical or pathological diagnosis (only for suspicious lesions confirmed pathologically) of cutaneous warts on the palmoplantar area by a dermatologist. The patients' ages range from 4 to 18 years old, and the number of warts must be a maximum of 20.

Exclusion Criteria: The exclusion criteria include pregnancy and breastfeeding, warts on the face, inguinal, and genital areas, hypersensitivity to topical vitamin D derivatives or fluorouracil, extensive warts requiring other treatments, and receiving any treatment in the past two months. Patients with confirmed immunodeficiency will also be excluded from the study.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Treatment respone | The number of lesions is recorded at 2 weeks, 4 weeks, and 8 weeks after the intervention.
  Treatment respone
  * No response: The wart shows no visible reduction in size, texture, or color, and there is no improvement in symptoms after the treatment.
  * Partial or Poor response: The wart demonstrates a reduction in size, texture, or color, but it is not completely resolved. Some improvement in symptoms may be noted, but the wart remains partially present.
  * Complete response: The wart is fully resolved with no visible signs remaining. All symptoms are eliminated, and the skin appears almost normal at the site of the wart.

SECONDARY OUTCOMES:
Number of Lesions | The number of lesions is recorded at 2 weeks, 4 weeks, and 8 weeks after the intervention.
  This outcome measures the total count of wart lesions present on a patient at each assessment point during the study. The number of lesions is recorded before the start of treatment and monitored at regular intervals throughout the treatment period and follow-up visits. The change in the number of lesions over time helps assess the effectiveness of the treatment in reducing wart lesions.
Size Change (Number of Lesions) | The size change is evaluated at 2 weeks, 4 weeks, and 8 weeks after the intervention.
  Size Change (Number of Lesions)
  This outcome tracks the change in size of the wart lesions over time, categorizing them into two options:
  * Decrease: The lesions have reduced in size compared to the initial measurement taken before the start of treatment.
  * Increase: The lesions have grown in size compared to the initial measurement taken before the start of treatment.
Adverse Events | Adverse events are assessed at 2 weeks, 4 weeks, and 8 weeks after the intervention.
  Adverse Events This outcome tracks the occurrence of any adverse events experienced by the patient during the study. Adverse events are monitored and recorded at each assessment point.
  * No: The patient does not experience any adverse events related to the treatment.
  * Yes: The patient experiences one or more adverse events. If "Yes," the adverse events are described in detail, including the type, severity, duration, and any measures taken to manage the events.
Photography | These photographs are taken at 0, 2 weeks, 4 weeks, and 8 weeks after the intervention.
  Photographs are taken of all patients at each assessment point to document the visual appearance of the wart lesions. This provides a visual record to support the assessment of treatment response and size change.

CONTACTS AND LOCATIONS:
Locations (1):
- Iran, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Undecided